CLINICAL TRIAL: NCT02309281
Title: Intravitreal Aflibercept (VEGF Trap-Eye) in Neovascular Age-related Macular Degeneration With Limited Response to Ranibizumab
Brief Title: Intravitreal Aflibercept in Neovascular AMD With Limited Response to Ranibizumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vista Klinik (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Dr. med. Katja Hatz, Prof., Vista Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eylea1
Record Dates: First submitted 2014-11-25; First posted 2014-12-05 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Eylea
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aflibercept 2mg (Other): Aflibercept 2mg (Eylea) is intravitreally applied. The first treatment interval with aflibercept will be 4 weeks and corresponding to the treat and extend regime intervals will be increased in 2-weeks-steps.
  Interventions: Drug: aflibercept 2mg

INTERVENTIONS:
Drug: aflibercept 2mg — Aflibercept 2mg (Eylea) is intravitreally applied. The first treatment interval with aflibercept will be 4 weeks and corresponding to the treat and extend regime intervals will be increased in 2-weeks-steps.
  Other Names: Eylea 2mg

SUMMARY:
Title: Intravitreal aflibercept (VEGF Trap-Eye) in neovascular age-related macular degeneration with limited response to ranibizumab

Purpose: The purpose of this investigator initiated study is to identify the duration of treatment effects of intravitreal aflibercept on sub- and intraretinal fluid and best corrected visual acuity (BCVA) in choroidal neovascularizations (CNV) due to age-related macular degeneration (AMD) in which the Optical coherence tomography (OCT) guided treatment interval failed to be extended to 6 weeks intervals in a treat and extend regimen.

Objectives: The primary objective is to evaluate the mean maximum recurrence-free treatment interval (Imax in weeks) with aflibercept treatment during the 24 months study peroid (for explanation see section Objectives). The individual maximum recurrence-free treatment interval (in weeks) at 24 weeks is defined as the maximum extension interval which is reached during the study follow-up period without showing any CNV activity (any intra-or subretinal fluid at OCT or new retinal hemorrhage). This measure reflects the duration of aflibercept effect in these lesions with limited response to ranibizumab. Key secondary Outcome Measures are mean changes in BCVA score at 24 weeks from baseline (Δ BCVAscore), mean changes in CRT (µm) at 24 weeks from baseline (Δ CRT), mean number of treatments needed during the 24 weeks study follow-up, number of participants with adverse events and serious adverse events (for further outcome measures see section Objectives).

Population: This outpatient study population will consist of a representative group of 33 male and female patients ≥ 50 years of age. The study population will include patients with subfoveal CNV secondary to AMD and being pre-treated with intravitreal ranibizumab in a treat and extend regimen and failed to be extended to 6-weeks intervals without showing CNV activity (for further information see section Criteria).

Interventions: 1-arm interventional study with 2mg aflibercept intravitreally up to 4-weekly. The first treatment interval with aflibercept will be 4 weeks and corresponding to the treat and extend regime intervals will be increased in 2-weeks-steps as long as no CNV activity (any intra-or subretinal fluid at OCT or new retinal hemorrhage) occurs. In case of occuring CNV activity the interval is shortened by 4 weeks with a minimum treatment interval of 4 weeks.

DETAILED DESCRIPTION:
Title of study: Intravitreal aflibercept (VEGF Trap-Eye) in neovascular age-related macular degeneration with limited response to ranibizumab

Study purpose: The purpose of this investigator initiated study is to identify the duration of treatment effects of intravitreal aflibercept (VEGF Trap-Eye) on sub- and intraretinal fluid and best corrected visual acuity (BCVA) in choroidal neovascularizations (CNV) due to age-related macular degeneration (AMD) in which the Optical coherence tomography (OCT) guided treatment interval failed to be extended to 6 weeks intervals in a treat and extend regimen.

Objectives: The primary objective is to evaluate the mean maximum recurrence-free treatment interval (Imax in weeks) with intravitreal aflibercept treatment in an OCT- and fundus examination- guided treat and extend regimen within a 24 weeks study period. The individual maximum recurrence-free treatment interval (in weeks) at 24 weeks is defined as the maximum extension interval which is reached during the study follow-up period without showing any CNV activity (any intra-or subretinal fluid at OCT or new retinal hemorrhage). This measure reflects the duration of aflibercept effect in these lesions with limited response to ranibizumab.

Secondary Objectives are:

* mean changes in BCVA score at 24 weeks compared to baseline (Δ BCVAscore=BCVAscore 24 weeks - BCVAscore Baseline)
* mean changes in CRT (central retinal thickness; in µm) at 24 weeks compared to baseline (Δ CRT=CRT 24 weeks - CRT Baseline)
* percentage of patients with a maximum recurrence-free treatment interval of more than 4 weeks at 24 weeks
* mean number of treatments needed during the 24 weeks study follow-up
* percentage of lesions showing incidence of fluorescein leakage at baseline and 24 weeks.
* mean change in total lesion area at 24 weeks compared to baseline (ΔTotalArea=TotalArea 24weeks - TotalArea Baseline)
* mean change in area of leakage from CNV at 24 weeks compared to baseline (ΔLeakageArea=LeakageArea 24weeks - LeakageArea Baseline)
* change of quality of life scores (VFQ-25, EQ 5D) from baseline to 24 weeks.
* number of participants with adverse events (not fullfilling the criteria of serious adverse events) as a measure of safety and tolerability of up to 4weekly dosing of aflibercept in CNV due to AMD
* number of participants with serious adverse events as a measure of safety and tolerability of up to 4weekly dosing of aflibercept in CNV due to AMD

Population: This outpatient study population will consist of a representative group of 33 male and female patients ≥ 50 years of age. The study population will include patients with predominantly classic, minimally classic, or occult lesions with no classic component, all with subfoveal CNV secondary to AMD. All patients are pre-treated with intravitreal ranibizumab in a treat and extend regimen and failed to be extended to 6-weeks intervals without showing CNV activity.

Inclusion criteria

* Male or female patients ≥ 50 years of age.
* Active subfoveal CNV secondary to AMD, including those with predominantly classic, minimally classic or occult lesions with no classic component.
* Pre-treatment with intravitreal ranibizumab in a treat and extend regimen with 2-weeks steps similar to the treat and extend regimen used in this study (see Study design) and failing to be extended to 6-weeks intervals without showing CNV activity (at least 2 attempts to extend from 4 to 6 weeks).
* Evidence that CNV extends under the geometric center of the foveal avascular zone.
* The total area of CNV (including all components) encompassed within the lesion must be ≥ 50% of the total lesion area.
* The total lesion area ≤ 12 disc areas for minimally classic or occult with no classic component and ≤ 9 disc areas (5400µm) in greatest linear dimension with predominantly classic lesions.
* BCVAscore of at least 23 letters (20/320) in the study eye using ETDRS charts.
* Willing and able to give written informed consent according to legal requirements, and have signed the consent form prior to initiation of any study procedure including withdrawal from exclusionary medications for the purpose of this study.
* Willing and able to comply with study procedures.

Exclusion criteria

* Subretinal hemorrhage in the study eye involving the center of the fovea, if the size of the hemorrhage is ≥ 50% of the total lesion area or ≥ 1 disc area.
* Presence of a retinal pigment epithelial tear or significant fibrosis involving the fovea in the study eye.
* Angioid streaks or precursors of CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, pathologic myopia.
* Concurrent disease in the study eye that could compromise visual acuity or require medical/surgical intervention during the study period.
* Vitreous hemorrhage or history of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye.
* Active intraocular inflammation in the study eye.
* Any active infection involving ocular adnexa including infectious conjunctivitis, keratitis, scleritis, endophthalmitis, as well as idiopathic or autoimmune-associated uveitis in either eye.
* History of uncontrolled glaucoma in the study eye (intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication).
* Aphakia with absence of the posterior capsule in the study eye.
* Prior treatment in the study eye with external-beam radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, transpupillary thermotherapy.
* History of submacular surgery or other surgical intervention for AMD in the study eye, glaucoma filtration surgery, corneal transplant surgery.
* Extraction of cataract with phacoemulsification within 3 months preceding Baseline, or a history of post-operative complications within the last 12 months preceding Baseline in the study eye.
* Use of other investigational drugs at the time of baseline, or within 30 days or 5 half- lives of baseline, whichever is longer (excluding vitamins + minerals).
* Previous violation of the posterior capsule in the study eye unless as a result of YAG posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation.
* History of other disease, metabolic dysfunction, examination finding, or clinical laboratory finding giving reasonable suspicion of a disease/condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications.
* Pregnant or nursing (lactating) women. Pregnancy is defined as the state after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/ml).
* History of hypersensitivity/allergy to fluorescein.
* Inability to obtain OCTs, fundus photographs, fluorescein angiograms of sufficient quality.

Study design/interventions: 1-arm interventional investigator-initiated study with 2mg aflibercept intravitreally with up to 4-weekly treatment in a treat and extend regimen. The first treatment interval with aflibercept will be 4 weeks and corresponding to the treat and extend regimen intervals will be increased in 2-weeks-steps as long as no CNV activity (any intra-or subretinal fluid at OCT or new retinal hemorrhage) occurs. In case of occuring CNV activity the interval is shortened by 4 weeks with a minimum treatment interval of 4 weeks. At every scheduled treat and extend visit (including baseline but excluding exit visit) an aflibercept injection is administered with a maximum of 6 injections during the study period.

Study visits: Baseline (4 weeks after last ranibizumab treatment), 4 weeks (28±2days), further visits according to treat and extend regimen (see above) at x weeks±2days with one week=7days, Exit visit (24 weeks±2days).

Study examinations/evaluations (both eyes):

* medical and ocular history (each visit)
* concomitant medication (each visit)
* adverse events (each visit and in between if necessary)
* BCVA score following ETDRS refraction protocol at 4m (each visit)
* SD-OCT scan (each visit)
* ophthalmic biomicroscopic examination including funduscopy (each visit)
* applanatory intraocular pressure measurement pre- and post injection (each visit)
* fluoresceine angiography (baseline and exit visit)
* quality of life questionaires VFQ-25 and EQ 5D (baseline and exit visit)

ELIGIBILITY:
Inclusion criteria

* Male or female patients ≥ 50 years of age.
* Active subfoveal CNV secondary to AMD, including those with predominantly classic, minimally classic or occult lesions with no classic component.
* Pre-treatment with intravitreal ranibizumab in a treat and extend regimen with 2-weeks steps similar to the treat and extend regimen used in this study (see Study design) and failing to be extended to 6-weeks intervals without showing CNV activity (at least 2 attempts to extend from 4 to 6 weeks).
* Evidence that CNV extends under the geometric center of the foveal avascular zone.
* The total area of CNV (including all components) encompassed within the lesion must be ≥ 50% of the total lesion area.
* The total lesion area ≤ 12 disc areas for minimally classic or occult with no classic component and ≤ 9 disc areas (5400µm) in greatest linear dimension with predominantly classic lesions.
* BCVAscore of at least 23 letters (20/320) in the study eye using ETDRS charts.
* Willing and able to give written informed consent according to legal requirements, and have signed the consent form prior to initiation of any study procedure including withdrawal from exclusionary medications for the purpose of this study.
* Willing and able to comply with study procedures.

Exclusion criteria

* Subretinal hemorrhage in the study eye involving the center of the fovea, if the size of the hemorrhage is ≥ 50% of the total lesion area or ≥ 1 disc area.
* Presence of a retinal pigment epithelial tear or significant fibrosis involving the fovea in the study eye.
* Angioid streaks or precursors of CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, pathologic myopia.
* Concurrent disease in the study eye that could compromise visual acuity or require medical/surgical intervention during the study period.
* Vitreous hemorrhage or history of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye.
* Active intraocular inflammation in the study eye.
* Any active infection involving ocular adnexa including infectious conjunctivitis, keratitis, scleritis, endophthalmitis, as well as idiopathic or autoimmune-associated uveitis in either eye.
* History of uncontrolled glaucoma in the study eye (intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication).
* Aphakia with absence of the posterior capsule in the study eye.
* Prior treatment in the study eye with external-beam radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, transpupillary thermotherapy.
* History of submacular surgery or other surgical intervention for AMD in the study eye, glaucoma filtration surgery, corneal transplant surgery.
* Extraction of cataract with phacoemulsification within 3 months preceding Baseline, or a history of post-operative complications within the last 12 months preceding Baseline in the study eye.
* Use of other investigational drugs at the time of baseline, or within 30 days or 5 half- lives of baseline, whichever is longer (excluding vitamins + minerals).
* Previous violation of the posterior capsule in the study eye unless as a result of YAG posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation.
* History of other disease, metabolic dysfunction, examination finding, or clinical laboratory finding giving reasonable suspicion of a disease/condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications.
* Pregnant or nursing (lactating) women. Pregnancy is defined as the state after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/ml).
* History of hypersensitivity/allergy to fluorescein.
* Inability to obtain OCTs, fundus photographs, fluorescein angiograms of sufficient quality.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
mean maximum recurrence-free treatment interval (Imax in weeks) with aflibercept treatment during the 24 months study peroid | 24 weeks
  All eligible patients have to show a maximum treatment interval with ranibizumab (pre-study period) of 4 weeks (failed to be extended to 6 weeks, see Inclusion criteria), meaning that the mean maximum treatment interval at baseline is 4 weeks. During the study the treatment intervals with aflibercept will be increased in 2-weeks steps corresponding to the treat and extend regime (see Study design). The individual maximum recurrence-free treatment interval (in weeks) at 24 weeks is defined as the maximum extension interval which is reached during the study follow-up period without showing any CNV activity (any intra-or subretinal fluid at OCT or new retinal hemorrhage). This measure reflects the duration of aflibercept effect in these lesions with limited response to ranibizumab.

SECONDARY OUTCOMES:
mean changes in BCVA score at 24 weeks compared to baseline (Δ BCVAscore=BCVAscore 24 weeks - BCVAscore Baseline) | 24 weeks
  changes in BCVA score from Baseline to 24weeks
mean changes in CRT (central retinal thickness; in µm) at 24 weeks compared to baseline (Δ CRT=CRT 24 weeks - CRT Baseline) | 24 weeks
  changes from the CRT from Baseline to 24weeks
percentage of patients with a maximum recurrence-free treatment interval of more than 4 weeks at 24 weeks | 24 weeks
  percentage of patients have to show a Maximum recurrence
mean number of treatments needed during the 24 weeks study follow-up | 24 weeks
  number of treatments needed during the 24 weeks study
percentage of lesions showing incidence of fluorescein leakage at baseline and 24 weeks. | 24 weeks
  percentage of lesions showing incidence of fluorescein leakage from baseline to week 24
mean change in total lesion area at 24 weeks compared to baseline (ΔTotalArea=TotalArea 24weeks - TotalArea Baseline) | 24 weeks
  changes in total lesion area from Baseline to 24weeks
mean change in area of leakage from CNV at 24 weeks compared to baseline (ΔLeakageArea=LeakageArea 24weeks - LeakageArea Baseline) | 24 weeks
  change in area of leakage from CNV from baseline to week 24
change of quality of life scores (VFQ-25, EQ 5D) from baseline to 24 weeks. | 24 weeks
  changes of VFQ-25 questionaire from Baseline to 24weeks
number of participants with adverse events (not fullfilling the criteria of serious adverse events) as a measure of safety and tolerability of up to 4weekly dosing of aflibercept in CNV due to AMD | 24 weeks
  number of AEs from Baseline to week 24
number of participants with serious adverse events as a measure of safety and tolerability of up to 4weekly dosing of aflibercept in CNV due to AMD | 24 weeks
  number of SAEs from Baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Katja Hatz, MD, Principal Investigator — Vista Klinik Binningen